CLINICAL TRIAL: NCT00786409
Title: Immunogenicity and Safety of the Quadrivalent HPV Vaccine Gardasil in Female Systemic Lupus Erythematosus Patients Aged 9-26
Brief Title: Immunogenicity and Safety of HPV Vaccine Gardasil in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15960A; MERCK: MISP for Gardasil#33598
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gardasil (Other): 30 patients will receive 0.5 ml Gardasil vaccine at months 0,2, and 6.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Gardasil — 0.5 ml Gardasil vaccine will be administered to each patient at months 0,2 and 6.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the HPV vaccine Gardasil in young women.

DETAILED DESCRIPTION:
Female patients with systemic lupus erythematosus (SLE) have been found have higher rates of persistent HPV infections and precancerous lesions compared to the healthy population. The HPV vaccine Gardasil has been found to be safe and efficacious in females aged 9 to 26 years. There are no data on the immunogenicity and safety of Gardasil in females with SLE. Immune dysfunction related to SLE itself and the immunosuppression secondary to treatment of SLE might prevent patients with SLE from developing an adequate immune response to the vaccine. Also, theoretically, the vaccine might induce a disease exacerbation or production of new autoantibodies.

The purpose of this study is to evaluate immunogenicity and safety of Gardasil and its effects on autoantibody profile in female SLE patients aged 9-26 years

ELIGIBILITY:
Inclusion Criteria:

* Age: 9 to 26 years of age
* Gender: Female
* All patients must fulfill the revised American College of Rheumatology Classification Criteria for SLE diagnosis.
* Current SLEDAI score ≤ 6
* Written, witnessed informed consent and/or assent will be obtained from the subject and the subject's parents (if under 18 years of age) or legally acceptable representative prior to enrollment

Exclusion Criteria:

* Acute exacerbation of disease within past 30 days which required increase in corticosteroid dose, initiation of a new immunosuppressive medication, or hospitalization
* Current SLEDAI score > 6
* Patients who have received rituximab in the last 6 months, or are currently on cyclophosphamide treatment
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine
* Previous administration of any HPV vaccine

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Wagner-Weiner, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Nath R, Mant C, Luxton J, Hughes G, Raju KS, Shepherd P, Cason J. High risk of human papillomavirus type 16 infections and of development of cervical squamous intraepithelial lesions in systemic lupus erythematosus patients. Arthritis Rheum. 2007 May 15;57(4):619-25. doi: 10.1002/art.22667. PMID 17471531

RESULTS

PARTICIPANT FLOW:
Groups:
- Gardasil Vaccine: 0.5 ml Gardasil vaccine at months 0, 2, and 6
Period: Overall Study
Arm/Group | Gardasil Vaccine
Started | 27
Completed | 20
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2
Not completed — Pregnancy | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: years] | 20.5 [12 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Anti-HPV 6 Seroconversion
Description: Percent Seropositive
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
percentage of participants | 93.8 [69.8 to 99.8]

2. Primary Outcome: Anti-HPV 6 GMT
Description: Geometric mean titre in milli-Merck units per ml (mMu/ml)
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Geometric Mean (95% Confidence Interval); unit: mMu/ml
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
mMu/ml | 427.0 [203.4 to 903.4]

3. Primary Outcome: Anti-HPV 11 Seroconversion
Description: % Seropositive
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

4. Primary Outcome: Anti-HPV 11 GMT
Description: Geometric mean titre in milli-Merck units per ml (mMu/ml)
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Geometric Mean (95% Confidence Interval); unit: mMu/ml
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
mMu/ml | 596.7 [303.6 to 1173.2]

5. Primary Outcome: Anti-HPV 16 Seroconversion
Description: % Seropositive
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

6. Primary Outcome: Anti-HPV 16 GMT
Description: Geometric mean titre in milli-Merck units per ml (mMu/ml)
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Geometric Mean (95% Confidence Interval); unit: mMu/ml
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
mMu/ml | 2263.2 [1019.3 to 5024.8]

7. Primary Outcome: Anti-HPV 18 Seroconversion
Description: % Seropositive
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
percentage of participants | 93.8 [69.8 to 99.8]

8. Primary Outcome: Anti-HPV 18 GMT
Description: Geometric mean titre in milli-Merck units per ml (mMu/ml)
Time Frame: 7 months
Population: 4 patients did not have month 7 samples available for analysis
Measure: Geometric Mean (95% Confidence Interval); unit: mMu/ml
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 16
mMu/ml | 331.9 [159.8 to 689.2]

9. Primary Outcome: SLEDAI Change Score
Description: Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): change from baseline to 7 months. The SLEDAI scale is a weighted sum of 16 clinical and 8 laboratory items. Scores range from 0 to 105 with higher scores indicating worse outcome. The variable analyzed here is the 7 month score minus the baseline score. Therefore negative values indicate an improvement in outcome.
Time Frame: 7 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 20
units on a scale | -1.65 [-2.85 to -0.44]

10. Secondary Outcome: Induction or Increase of Autoantibodies (Conversion From Negative Anti-RNP to Positive Anti-RNP) Anti-RNP
Time Frame: 7 months
Population: 8 patients were negative for anti-RNP at entry
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 8
Participants | 0

11. Secondary Outcome: Induction or Increase of Autoantibodies (Conversion From Negative Smith to Positive Smith)
Time Frame: 7 months
Population: 13 patients were Smith negative at entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 13
Participants | 0

12. Secondary Outcome: Induction or Increase of Autoantibodies (Conversion From Lupus Anticoagulant Negative to Lupus Anticoagulant Positive)
Time Frame: 7 months
Population: 17 patients were Lupus anticoagulant negative at entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 17
Participants | 2

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Gardasil Vaccine
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gardasil Vaccine (N=27)
Progression of Class IV Nephritis to Renal Failure (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gardasil Vaccine (N=27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes